CLINICAL TRIAL: NCT00394628
Title: A Phase 1b/2a, Multicenter, Open-Label Study of AQ4N in Combination With Radiation Therapy and Temozolomide, to Evaluate the Safety, Tolerability, and Efficacy in Subjects With Newly Diagnosed Glioblastoma Multiforme
Brief Title: AQ4N in Combination With Radiotherapy and Temozolomide in Subjects With Newly Diagnosed Glioblastoma Multiforme
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Novacea (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 021-003
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2007-05-30 (Estimated); Status verified 2007-05

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme; Radiotherapy; temozolomide; adjuvant temozolomide
MeSH Terms: conditions — Glioblastoma | interventions — AQ4N; Temozolomide; Radiotherapy

INTERVENTIONS:
Drug: AQ4N
Drug: Temozolomide
Procedure: Radiotherapy

SUMMARY:
Phase 1b of the study, will evaluate the safety and tolerability of AQ4N treatment at three different dose levels.

Phase 2a of the study, will further evaluate the safety, tolerability, and in addition efficacy of AQ4N treatment at a tolerated dose selected from Phase 1b.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven intracranial Glioblastoma Multiforme (GBM) with diagnosis established by biopsy or resection within 5 weeks prior to enrollment.
* Cranial MRI or contrast CT performed 14 days prior to study entry. Subjects without measurable or assessable disease are eligible.
* Plan to begin partial brain radiotherapy within 24-72 hours after beginning AQ4N, and within 35 days (5 weeks) of the surgery, or if surgery cannot be performed, the biopsy that confirms GBM diagnosis. Radiation therapy must be given by external beam to a partial brian field in daily fractions of 2.0 Gy, to a planned total dose to the tumor of 60.0 Gy over 6 weeks.
* Age equal to or greater than 18 years and life expectancy > 10 weeks.
* Karnofsky performance status of > 60.
* Adequate bone marrow, liver and renal functions (tests must be performed within 14 days prior to enrollment).
* Negative serum or urine pregnancy test (females of childbearing potential only).
* Willingness to use effective contraception (both males and females of child-bearing potential) throughout the study and for at least 2 months after study treatment.
* Able and willing to give informed consent.

Exclusion Criteria:

* Previous radiotherapy to the brain.
* Previous cytotoxic drug therapy, non-cytotoxic drug therapy, or experimental drug therapy directed against the brain tumor. Subjects who received Gliadel wafers will be excluded.
* Subjects previously treated with enzyme-induced antiepileptic drugs (EIAEDs) must have discontinued treatment with these agent(s) greater than or equal to 2 weeks prior to enrollment.
* A history of any other primary malignancy that has not been treated with curative intent and that has not been in complete remission for at least 2 years (exempt from the two year limit are non-melanoma skin cancer and cervical carcinoma in-situ on biopsy or a squamous intraepithelial lesion on PAP smear).
* Active infection.
* Any significant medical illnesses or toxicities that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the subjects' ability to tolerate this therapy. Subjects must not have any disease that will obscure toxicity or dangerously alter drug metabolism, e.g. congestive heart failure, moderate to severe liver and renal disease, other cancers.
* Cardiac ejection fraction (LVEF) by multiple gated acquisition scan (MUGA) less than the institutional lower limit of normal.
* Prior investigational therapy within the past 28 days.
* Prior AQ4N therapy.
* Hypersensitivity to AQ4N or to any ingredients contained in the drug formulation.
* Hypersensitivity to temozolomide or to any ingredients contained in the drug formulation and dacarbazine (DTIC).
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-10

PRIMARY OUTCOMES:
Phase 1b: Evaluation of the safety and tolerability of AQ4N in combination with radiation therapy and temozolomide (TEMODAR®)for the treatment of glioblastoma multiforme (GBM). Dose levels for the Phase 2a will be selected.
Phase 2a: Rate of progression-free survival at 6 months.

SECONDARY OUTCOMES:
Phase 2a: Rate of progression-free survival at 12 months
Percent of subjects alive at 12 months
Duration of progression-free survival
Time to progression
Duration of overall survival

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California, Los Angeles, Los Angeles, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Henry Ford Health Systems, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Baylor Research Institute, Dallas, Texas